CLINICAL TRIAL: NCT02201238
Title: A Pharmacokinetics Study Comparing Systemic Exposure of Topical Diclofenac/Menthol Gels Versus Voltaren Gel and Oral Diclofenac Sodium in Healthy Volunteers at Steady State
Brief Title: Pharmacokinetics Study Comparing Topical Diclofenac/Menthol Gels With Voltaren Gel and Oral Diclofenac Sodium
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 202188; RH02175 (Other: GSK)
Record Dates: First submitted 2014-07-24; First posted 2014-07-28 (Estimated); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Diclofenac; Menthol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Diclofenac sodium/menthol gel (in tube) (Experimental): 1% diclofenac sodium plus 3% menthol gel (in 30g aluminium tube). Dose given- 4g applied topically to a 400cm2 (20cm x 20cm) area of the skin, four times daily for three consecutive days with 5h between adjacent doses on the same day
  Interventions: Drug: Diclofenac sodium; Drug: Menthol
- Diclofenac sodium/menthol gel (in roll-on device) (Experimental): 1% diclofenac sodium plus 3% menthol gel (in roll-on applicator device supplied in 30g plastic bottles). Dose given- 4g applied topically to a 400cm2 (20cm x 20cm) area of the skin, four times daily for three consecutive days with 5h between adjacent doses on the same day
  Interventions: Drug: Diclofenac sodium; Drug: Menthol
- Diclofenac sodium tablets (Active Comparator): 50mg diclofenac sodium tablets administered orally, three times daily for three consecutive days with 6h between adjacent doses on the same day
  Interventions: Drug: Diclofenac sodium
- Voltaren gel (Active Comparator): Voltaren gel supplied in 100g aluminium tube. Dose given- 4g applied topically to a 400cm2 (20cm x 20cm) area of the skin, four times daily for three consecutive days with 5h between adjacent doses on the same day
  Interventions: Drug: Diclofenac sodium

INTERVENTIONS:
Drug: Diclofenac sodium — Diclofenac sodium
Drug: Menthol — Menthol
  Arms: Diclofenac sodium/menthol gel (in roll-on device); Diclofenac sodium/menthol gel (in tube)

SUMMARY:
This research study is being conducted to characterize the pharmacokinetic properties of a new topical medication (MFC51123) that contains two active ingredients (diclofenac and menthol) in two formulation packages. One formulation package is in the form of a gel in aluminum tube and the other one in the form of a gel in roll-on applicator bottle. Additionally, as a comparison, the pharmacokinetic properties of a marketed diclofenac gel and an oral diclofenac treatment will also be characterized. This topical diclofenac/menthol gel has being developed to treat mild to moderate pain and inflammation, such as acute sport injuries, sprains and strains. The rationale for conducting the study is to prove that repeated topical treatment of the new diclofenac + menthol formulation in either of the two packages does not result in unsafe systemic exposure.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 to 50 years
* Body mass index between 19-28 (kg/m2)

Exclusion Criteria:

* Pregnant or lactating females
* Participants having intolerance or hypersensitivity to study material
* Participants having positive results for HIV, Hepatitis B or Hepatitis C
* Participants having skin lesion at site of application
* Participants having history of alcohol or drug abuse

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2014-11-21 (Actual); Study Completion 2014-11-21 (Actual)

PRIMARY OUTCOMES:
AUC48-72 hrs of Diclofenac gel in tube/AUC48-72 hrs of oral Diclofenac | 20 days
  Ratio of area under the plasma concentration time curve from 48-72 hrs (AUC48-72 hrs) of Diclofenac gel in tube and AUC48-72 hrs of oral Diclofenac during the final 24 hours of dosing at steady state will assess systemic exposure to Diclofenac from gel as compared to that from oral Diclofenac
Cmax of Diclofenac gel in tube/Cmax of oral Diclofenac | 20 days
  Ratio of maximum plasma concentration (Cmax) of Diclofenac gel in tube and Cmax of oral Diclofenac during the final 24 hours of dosing at steady state will assess systemic exposure to Diclofenac from gel as compared to that from oral Diclofenac
AUC48-72 hrs of Diclofenac gel in roll-on device/AUC48-72 hrs of oral Diclofenac | 20 days
  Ratio of AUC48-72 hrs of Diclofenac gel in roll-on device and AUC48-72 hrs of oral Diclofenac during the final 24 hours of dosing at steady state will assess systemic exposure to Diclofenac from roll-on device as compared to that from oral Diclofenac
Cmax of Diclofenac gel in roll-on device/Cmax of oral Diclofenac | 20 days
  Ratio of Cmax of Diclofenac gel in roll-on device and Cmax of oral Diclofenac during the final 24 hours of dosing at steady state will assess systemic exposure to Diclofenac from roll-on device as compared to that from oral Diclofenac

SECONDARY OUTCOMES:
Cmin of Diclofenac gel in tube/Cmin of oral Diclofenac | 20 days
  Ratio of minimum plasma concentration (Cmin) of Diclofenac gel in tube and Cmin of oral Diclofenac during the final 24 hours of dosing at steady state will assess systemic exposure to Diclofenac from gel as compared to that from oral Diclofenac
Tmax of Diclofenac gel in tube/Tmax of oral Diclofenac | 20 days
  Ratio of time to maximum plasma concentration (Tmax) of Diclofenac gel in tube and Tmax of oral Diclofenac during the final 24 hours of dosing at steady state will assess systemic exposure to Diclofenac from gel as compared to that from oral Diclofenac
Cmin of Diclofenac gel in roll-on device/Cmin of oral Diclofenac | 20 days
  Ratio of Cmin of Diclofenac gel in roll-on device and Cmin of oral Diclofenac during the final 24 hours of dosing at steady state will assess systemic exposure to Diclofenac from roll-on device as compared to that from oral Diclofenac
Tmax of Diclofenac gel in roll-on device/Tmax of oral Diclofenac | 20 days
  Ratio of Tmax of Diclofenac gel in roll-on device and Tmax of oral Diclofenac during the final 24 hours of dosing at steady state will assess systemic exposure to Diclofenac from roll-on device as compared to that from oral Diclofenac
Cmax of Diclofenac gel in tube/Cmax of Diclofenac in Voltaren gel | 20 days
  Ratio of Cmax of Diclofenac gel in tube and Cmax of Voltaren gel during the final 24 hours of dosing at steady state will assess systemic exposure to Diclofenac from gel as compared to that from Voltaren gel
Cmax of Diclofenac gel in roll-on device/Cmax of Diclofenac in Voltaren gel | 20 days
  Ratio of Cmax of Diclofenac gel in roll-on device and Cmax of Voltaren gel during the final 24 hours of dosing at steady state will assess systemic exposure to Diclofenac from roll-on device as compared to that from Voltaren gel
Cmin of Diclofenac gel in tube/Cmin of Diclofenac in Voltaren gel | 20 days
  Ratio of Cmin of Diclofenac gel in tube and Cmin of Voltaren gel during the final 24 hours of dosing at steady state will assess systemic exposure to Diclofenac from gel as compared to that from Voltaren gel
Cmin of Diclofenac gel in roll-on device/Cmin of Diclofenac in Voltaren gel | 20 days
  Ratio of Cmin of Diclofenac gel in roll-on device and Cmin of Voltaren gel during the final 24 hours of dosing at steady state will assess systemic exposure to Diclofenac from roll-on device as compared to that from Voltaren gel
AUC48-72 hrs of Diclofenac gel in tube/AUC48-72 hrs of Diclofenac in Voltaren gel | 20 days
  Ratio of AUC48-72 hrs of Diclofenac gel in tube and AUC48-72 hrs of Voltaren gel during the final 24 hours of dosing at steady state will assess systemic exposure to Diclofenac from gel as compared to that from Voltaren gel
AUC48-72 hrs of Diclofenac gel in roll-on device/AUC48-72 hrs of Diclofenac in Voltaren gel | 20 days
  Ratio of AUC48-72 hrs of Diclofenac gel in roll-on device and AUC48-72 hrs of Voltaren gel during the final 24 hours of dosing at steady state will assess systemic exposure to Diclofenac from roll-on device as compared to that from Voltaren gel
Tmax of Diclofenac gel in tube/Tmax of Diclofenac in Voltaren gel | 20 days
  Ratio of Tmax of Diclofenac gel in tube and Tmax of Voltaren during the final 24 hours of dosing at steady state will assess systemic exposure to Diclofenac from gel as compared to that from Voltaren gel
Tmax of Diclofenac gel in roll-on device/Tmax of Diclofenac in Voltaren gel | 20 days
  Ratio of Tmax of Diclofenac gel in roll-on device and Tmax of Voltaren during the final 24 hours of dosing at steady state will assess systemic exposure to Diclofenac from roll-on device as compared to that from Voltaren gel
Cmax of Menthol in gel/Cmax of Menthol reported in literature | 20 days
  Ratio of Cmax of Menthol in tube and Cmax of Menthol reported in literature will assess systemic exposure to menthol from gel tube as compared to that reported in literature
Cmax of Menthol in roll-on device/Cmax of Menthol reported in literature | 20 days
  Ratio of Cmax of Menthol in roll-on device and Cmax of Menthol reported in literature will assess systemic exposure of menthol from roll-on device as compared to that reported in literature
Cmin of Menthol in gel/Cmin of Menthol reported in literature | 20 days
  Ratio of Cmin of Menthol in tube and Cmin of Menthol reported in literature will assess systemic exposure to menthol from gel tube as compared to that reported in literature
Cmin of Menthol in roll-on device/Cmin of Menthol reported in literature | 20 days
  Ratio of Cmin of Menthol in roll-on device and Cmin of Menthol reported in literature will assess systemic exposure of menthol from roll-on device as compared to that reported in literature
Tmax of Menthol in gel/Tmax of Menthol reported in literature | 20 days
  Ratio of Tmax of Menthol in tube and Tmax of Menthol reported in literature will assess systemic exposure to menthol from gel tube as compared to that reported in literature
Tmax of Menthol in roll-on device/Tmax of Menthol reported in literature | 20 days
  Ratio of Tmax of Menthol in roll-on device and Tmax of Menthol reported in literature will assess systemic exposure of menthol from roll-on device as compared to that reported in literature
T1/2 of Menthol in gel/T1/2 of Menthol reported in literature | 20 days
  Ratio of half time elimination (T1/2) of Menthol in tube and T1/2 of Menthol reported in literature will assess systemic exposure to menthol from gel tube as compared to that reporetd in literature
T1/2 of Menthol in roll-on device/T1/2 of Menthol reported in literature | 20 days
  Ratio of T1/2 of Menthol in roll-on device and T1/2 of Menthol reported in literature will assess systemic exposure of menthol from roll-on device as compared to that reported in literature
AUC48-72 hrs of Menthol in gel/AUC48-72 hrs of Menthol reported in literature | 20 days
  Ratio of AUC48-72 hrs of Menthol in gel and AUC48-72 hrs of Menthol reported in literature will assess systemic exposure to menthol from gel tube as compared to that reported in literature
AUC48-72 hrs of Menthol in roll-on device/AUC48-72 hrs of Menthol reported in literature | 20 days
  Ratio of AUC48-72 hrs of Menthol in roll-on device and AUC48-72 hrs of Menthol reported in literature will assess systemic exposure of menthol from roll-on device as compared to that reported in literature
AUC48-72 hrs of Voltaren gel/AUC48-72 hrs of oral Diclofenac | 20 days
  Ratio of AUC48-72 hrs of Voltaren gel and AUC48-72 hrs of oral Diclofenac will assess systemic exposure of Voltaren gel as compared to oral Diclofenac
Cmax of Voltaren gel/Cmax of oral Diclofenac | 20 days
  Ratio of Cmax of Voltaren gel and Cmax of oral Diclofenac will assess systemic exposure of Voltaren gel as compared to oral Diclofenac
T1/2 of Diclofenac gel in tube/T1/2 of oral Diclofenac | 20 days
  Ratio of T1/2 of Diclofenac gel in tube and T1/2 of oral Diclofenac will assess systemic exposure to Diclofenac from gel as compared to that from oral Diclofenac
T1/2 of Diclofenac gel in roll-on device/T1/2 of oral Diclofenac | 20 days
  Ratio of T1/2 of Diclofenac gel in roll-on device and T1/2 of oral Diclofenac will assess systemic exposure to Diclofenac from roll-on device as compared to that from oral Diclofenac
T1/2 of Diclofenac gel in tube/T1/2 of Diclofenac in Voltaren gel | 20 days
  Ratio of T1/2 of Diclofenac gel in tube and T1/2 of Voltaren gel will assess systemic exposure to Diclofenac from gel tube as compared to that from Voltaren gel
T1/2 of Diclofenac gel in roll-on device/T1/2 of Diclofenac in Voltaren gel | 20 days
  Ratio of T1/2 of Diclofenac gel in roll-on device and T1/2 of Voltaren gel will assess systemic exposure to Diclofenac from roll-on device as compared to that from Voltaren gel
Adverse event monitoring | 27 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Buffalo, New York, United States

REFERENCES:
- See also: Results for the study 202188 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/202188?search=study&search_terms=202188#rs